CLINICAL TRIAL: NCT06242886
Title: The Effect of Oxytocin Massage After Caesarean Section on Anthropometric Characteristics of the Newborn and Breastfeeding Self-Efficacy: A Single Blind, Randomized Controlled Study
Brief Title: After Caesarean Section Oxitocin Breast Massage Anthropometric Characteristics of the Newborn
Acronym: OM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Massage
Record Dates: First submitted 2024-01-12; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Breastfeeding, Exclusive; Breastfeeding
Keywords: Breastfeeding self-efficacy; C-section,; oxytocin
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Intervention Model Description: A Single Blind, Randomized Controlled Study
Who Masked: Investigator, Outcomes Assessor
Masking Description: The mothers included in the study were blind to each other in terms of application, and the researcher who collected the data was blind to the groups in the study in terms of analysis and reporting. Breast and oxytocin massage and follow-up were carried out by the researcher (FŞB), who could not be blind to the applications. Randomization was done by another researcher (AYK). To avoid bias, the researcher who commissioned the study (FŞB) was not involved in any step of the data collection and statistical evaluation process
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Oxytocin massage (Experimental): The mother was positioned on a chair with her breasts bare and free, placing her arms on the table at her height and her head on her arms. The researcher who applied the massage applied the massage up and down to either side of the spine between the mother's scapula bones with her thumbs in front and pressing her fists tightly and making small circular movements with her thumbs for three minutes. The mothers received four oxytocin massages over the course of 24 hours.
  Interventions: Behavioral: Oxytocin massage
- Breast massage (Experimental): The mother's upper clothes were removed by the researcher. With the palms of the hand the breast grasped from the bottom and top. The hands were advanced by pressing slowly from the base of the nipple towards the nipple. With the palms, the breast was grasped from the bottom and top and gently pressed. Using fingertips, the breast was scanned by massaging from the base of the nipple to the nipple in circular movements. The mothers received breast massage four times over the course of 24 hours.
  Interventions: Behavioral: and Breast massage
- Control (No Intervention): No intervention

INTERVENTIONS:
Behavioral: Oxytocin massage — Oxytocin massage group: The mother was positioned on a chair with her breasts bare and free, placing her arms on the table at her height and her head on her arms. The researcher who applied the massage applied the massage up and down to either side of the spine between the mother's scapula bones with her thumbs in front and pressing her fists tightly and making small circular movements with her thumbs for three minutes. The mothers received four oxytocin massages over the course of 24 hours.
  Arms: Oxytocin massage
Behavioral: and Breast massage — Breast massage group: The mother's upper clothes were removed by the researcher. With the palms of the hand the breast grasped from the bottom and top. The hands were advanced by pressing slowly from the base of the nipple towards the nipple. With the palms, the breast was grasped from the bottom and top and gently pressed. Using fingertips, the breast was scanned by massaging from the base of the nipple to the nipple in circular movements. The mothers received breast massage four times over the course of 24 hours.
  Arms: Breast massage

SUMMARY:
Background: Delays in breastfeeding and milk release after cesarean section may negatively affect the early initiation of breastfeeding and the mother's breastfeeding self-efficacy.

Research Aims: The aim of this study was to investigate the effect of breast and oxytocin massage after cesarean section on the anthropometric characteristics of the newborn and breastfeeding self-efficacy.

Methods: The study was conducted in a single-blind randomized controlled type and 126 mothers who delivered by cesarean section in the postpartum department of a private hospital in Istanbul/Turkey were randomized into three groups as 42 breast massage, 42 oxytocin massage and 42 control group.

DETAILED DESCRIPTION:
Background: Delays in breastfeeding and milk release after cesarean section may negatively affect the early initiation of breastfeeding and the mother's breastfeeding self-efficacy.

Research Aims: The aim of this study was to investigate the effect of breast and oxytocin massage after cesarean section on the anthropometric characteristics of the newborn and breastfeeding self-efficacy.

Methods: The study was conducted in a single-blind randomized controlled type and 126 mothers who delivered by cesarean section in the postpartum department of a private hospital in Istanbul/Turkey were randomized into three groups as 42 breast massage, 42 oxytocin massage and 42 control group.

Mothers who had a cesarean delivery and were in the first 24 hours after birth were divided into three separate groups: breast massage, oxytocin massage and control group. Data Collection Form, LACTH, Infant Follow-up Form and Breastfeeding Self-Efficacy Scale were applied to all mothers included in the sampling in the postpartum period.

Oxytocin massage group: The mother was positioned on a chair with her breasts bare and free, placing her arms on the table at her height and her head on her arms. The researcher who applied the massage applied the massage up and down to either side of the spine between the mother's scapula bones with her thumbs in front and pressing her fists tightly and making small circular movements with her thumbs for three minutes. The mothers received four oxytocin massages over the course of 24 hours.

Breast massage group: The mother's upper clothes were removed by the researcher. With the palms of the hand the breast grasped from the bottom and top. The hands were advanced by pressing slowly from the base of the nipple towards the nipple. With the palms, the breast was grasped from the bottom and top and gently pressed. Using fingertips, the breast was scanned by massaging from the base of the nipple to the nipple in circular movements. The mothers received breast massage four times over the course of 24 hours.

Control group: Mothers were discontinued from routine care at the clinic.

ELIGIBILITY:
Inclusion Criteria:

* The study included mothers between the ages of 18 and 35, who were primiparous, due (37-42 GW) and cesarean section, who could understand and speak Turkish, who had no anatomical problems with their breasts, and who were in the first 24 hours after birth.

Exclusion Criteria:

* Mothers with communication problems, having a chronic illness, breastfeeding related problems (breast or newborn) and mothers with newborns with IUGR or genetic disease were not included in the study.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Postpartum, primiparous woman
Enrollment: 42 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-08-20 (Actual); Study Completion 2023-09-20 (Actual)

PRIMARY OUTCOMES:
Breastfeeding Self-Efficacy | Three times=immediately after birth, the first 24 hours after birth, and the 7th day after birth
  Breastfeeding Self-Efficacy Scale Total Score; Breastfeeding Charting System (LATCH) Turkish validity and reliability were made by Yenal and Okumuş [12]. Scale was developed to evaluate the breastfeeding. On the LATCH scale, a score of 0, 1 or 2 is given for each criterion. A minimum of 0-Maximum score of 10 points is taken from the scale. A low score by the mother indicates that she needs help with breastfeeding. Scoring is done by observing breastfeeding.
Breastfeeding success | Three times= immediately after birth, the first 24 hours after birth, and the 7th day after birth
  Breastfeeding success (LATCH) total score; As the LATCH score increases, it is understood that breastfeeding success is high. LATCH Cronbach's Alpha value: It was found to be 0.95 by Yenal and Okumuş [12]. In this study, 0.86 found. Developed to evaluate the breastfeeding self-efficacy levels of mothers. The Breastfeeding Self-Efficacy Short Form Scale is a Likert-type scale with 5 points. The minimum score that can be taken from the scale is 14 and the maximum score is 70. The higher the score, the higher the breastfeeding shows self-efficacy. The Turkish validity and reliability study of the scale was conducted by Tokat et al.[13] and Cronbach's Alpha value was found to be 0.86
Newborn Anthropometric Characteristics | Three times= immediately after birth, the first 24 hours after birth, and the 7th day after birth
  Weight

CONTACTS AND LOCATIONS:
Locations (1):
- Fatma Şule Bilgiç, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided